CLINICAL TRIAL: NCT05487742
Title: Evaluation of Neuroprotective Effect of Dexmedetomidine in Traumatic Brain Injury
Brief Title: Neuroprotective Effect of Dexomitomidine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Wafaa Madhy Atia Abdelwahed, lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 35526/6/22
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Dexmedetomidine Neuroprotective Effect in Traumatic Brain Injury
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: no participant ,investigator or outcome assessor in ICU know in which group patient is allocated
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (control group): (Placebo Comparator): Patients of this group receive placebo infusion for 72 hours.
  Interventions: Drug: placebo salin infusion
- Group II (DEX group): (Active Comparator): Patients of this group receive 0.5 ug/kg/hr dexmedetomidine continuous infusion for 72 hour
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine will be infused for 72 hour in mild and moderate traumatic brain injury patient
  Arms: Group II (DEX group):
Drug: placebo salin infusion — salin infused as aplacebo for 72 hours
  Arms: Group I (control group):

SUMMARY:
patient wih mild to moderate traumatic brain injury in ICU will be randomisly distributed into two groups Group I (control group): Patients of this group receive placebo infusion for 72 hours. Group II (DEX group): Patients of this group receive 0.5 ug/kg/hr dexmedetomidine continuous infusion for 72 hour Patient demographics, including age, sex, weight, primary diagnosis, Acute Physiology and Chronic Health Evaluation (APACHE) II score and postresuscitation Glasgow Coma Scale (GCS) score will be collected. CBF will be measured at pre-sedation and after cessation of sedation (dexmedetomidine administration). The CMRe and CMRe/CBF will also be calculated. Measurements of blood gas analysis and haemodynamic parameters [systolic blood pressure (SBP), diastolic blood pressure (DBP), MAP and heart rate (HR)] will be collected at pre-sedation and after cessation of sedation (dexmedetomidine administration).

DETAILED DESCRIPTION:
Assessment will be done for the patients by taking careful medical history for any medical disorder, therapeutic anticoagulant, allergy to chemical compounds or addiction problems, and performing trauma survey check up ( chest x-ray, abdomen US, CT brain for documentation of injury) with general and physical examination for CNS (assessement of GCS) , chest, heart, abdomen and peripheral limbs for any abnormality . Then, routine and relative investigations will be carried out such as complete blood picture, renal and liver function tests, coagulation tests and random blood sugar.

all patients will be monitored with five- lead ECG, non-invasive blood pressure, pulse oximetry and end tidal CO2. Then a 20 gauge IV cannula will be inserted into a peripheral upper extremity vein for drug administration and ( DEX group) patients received 0.5 ug /kg/hr dexmedetomidine continuous infusion for 72 hour. Ephedrine will be administrated to maintain the MAP at the pre-sedation level if BP decrease 20 % from baseline BP and atropine if pulse decrease below 50 b/m . No extra sedatives, other vasoactive drugs or volume resuscitation will be used during sedation. Patient demographics, including age, sex, weight, primary diagnosis, Acute Physiology and Chronic Health Evaluation (APACHE) II score and postresuscitation Glasgow Coma Scale (GCS) score will be collected. CBF will be measured at pre-sedation and after cessation of sedation (dexmedetomidine administration). The CMRe and CMRe/CBF will also be calculated. Measurements of blood gas analysis and haemodynamic parameters [systolic blood pressure (SBP), diastolic blood pressure (DBP), MAP and heart rate (HR)] will be collected at pre-sedation and after cessation of sedation (dexmedetomidine administration).

CBF measurement :

CBF will be evaluated in the extra-cranial internal carotid artery (ICA) and vertebral artery (VA) using a spectral Doppler ultrasound technique . Briefly, the procedure will be performed with the patient in the supine position with a 7.5-MHz linear array transducer of a colour coded ultrasound system . The patients' head will slightly be elevated and turned to the contralateral side at a 25 - 40 angle for ICA measurements and at a 10 angle for VA measurements. ICA will be assessed at the segment located 1.5 cm distal to the carotid bifurcation and VA will be measured between the transverse processes of the C4 and C5 vertebrae.

Blood flow velocities will be obtained by keeping the Doppler insonation angle at a standard 60. Time averaged flow velocity (TAV) will be determined as the integral of the mean flow velocities of all moving particles passing the sample volume over 3-5 complete cardiac cycles. The TAV, peak systolic velocity, end-diastolic velocity and inner vessel diameter (d) will be measured during the bilateral ICA and VA CBF measurements. The intravascular flow volume (FV) of each artery will be calculated by the formula: FV= TAV x (d/2) x ℼ CBF will be calculated as the sum of bilateral ICA and VA flow volumes. All ultrasound examinations will be performed in triplicate by the same radiologist using the same Doppler ultrasonography device.

CBF reduction will be calculated as:

(pre-sedation CBF - during-sedation CBF) / pre-sedation CBF x100.

CMRe evaluation :

An 18-gauge venous catheter (Arrow International Inc., Bernville, PA) will be introduced into the right internal jugular vein at the level of the cricothyroid membrane and passed into the jugular bulb or at the base of the skull in a retrograde fashion with ultrasound guidance, as previously described [12]. Blood samples for jugular venous oxygen saturation (SjvO2) measurements will be collected intermittently by aspiration at a rate of less than 1.5 ml min . Arterial oxygen saturation (SaO2) and partial pressure of carbon dioxide (PaCO2) were assessed in blood samples taken from the femoral artery. The CMRe and oxygen extraction ratio (OER) were calculated as follows:

CMRe = CBFx (SaO2ml_1 _ SjvO2ml_1) (relative units):

OER = (SaO2 _ SjvO2)/SaO2 The CMRe / CBF ratio was also determined at each time point. The reduction in CMRe was calculated using the method described above. 80 Patients will be randomly classified using sealed envelope into two equal groups each of 40 patients Group I (control group): Patients of this group receive placebo infusion for 72 hours. Group II (DEX group): Patients of this group receive 0.5 ug/kg/hr dexmedetomidine continuous infusion for 72 hour

ELIGIBILITY:
1. Patients of either sex
2. Age ranged from 18-60 years
3. Patients with mild to moderate traumatic brain injury assessed by CT and 8< GCS < 15 -

Exclusion Criteria:

1 - Patient relative refusal. 2-Severe traumatic brain injury GCS < 8 3-prescence of other organ injury. 4-MAP lower than 80 mmHg 5- hepatic or kidney function dysfunction 6-received any vasoactive agents or sedatives or recieve drugs that affect CBF during the experiment 7- Pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The change in CBF during sedation. | 6 months
  cerebral blood flow will be measured whether changed by dexmedetomine infusion or not

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta University, Tanta, Egypt